CLINICAL TRIAL: NCT04130412
Title: Open Versus Arthroscopic Release for Lateral Patellar Compression Syndrome: Comparative Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hawler Medical University (Other)
Responsible Party: Principal Investigator, Sherwan Ahmed Ali Hamawandi, Assistant professor of orthopedic surgery, Hawler Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HMU/Sherwan5
Record Dates: First submitted 2019-10-13; First posted 2019-10-17 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-06

CONDITIONS: Knee Arthroscopy
Keywords: Lateral patellar compression syndrome; Arthroscopic release; Open release
MeSH Terms: interventions — Joint Capsule Release

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Open release of lateral retinaculae (Active Comparator): This group was treated by open release of lateral retinaculae after diagnosis of lateral compression syndrome by arthroscopy
  Interventions: Procedure: open release
- Arthroscopic release of lateral retinaculae (Active Comparator): This group was treated by arthroscopic release
  Interventions: Procedure: open release

INTERVENTIONS:
Procedure: open release — Open release of lateral retinaculae
  Other Names: Arthroscopic release

SUMMARY:
Chronic anterior knee pain with a stable patella is often associated with overload and increased pressure on the lateral facet due to pathologic lateral soft-tissue restraints. "Lateral pressure in flexion" is a term describing the pathologic process of increasing contact pressure over the lateral patellar facet as knee flexion progresses. Eighty patients were involved in this study, and it was divided into 2 random groups; Group A (40 patients)(odd number) were treated with open release after diagnostic arthroscopy and Group B (40 patients)(even number) were treated by arthroscopic release. All these patients are diagnosed as lateral patellar compression syndrome depending on clinical features, MRI and diagnostic arthroscopy. All patients were followed by Lysholm knee scaling score before surgery and two weeks , six weeks then 6 months after surgery.

DETAILED DESCRIPTION:
This study was done by two orthopedic surgeons working in three hospitals from March 2016 to April 2018, Eighty patients were involved in this study, and it was divided into 2 matched groups; Group A (40 patients) were treated with open release after diagnostic arthroscopy and Group B (40 patients) were treated by arthroscopic release. All these patients are diagnosed as lateral patellar compression syndrome depending on clinical features, MRI ( figure 1)and diagnostic arthroscopy. All patients were followed by Lysol knee scaling score before surgery , two weeks , six weeks then 6 months after surgery. The two groups are matched related to age and gender. 52 patients are females and age ranged from 21-48 years.

Exclusion criteria are 1. Smoking 2.Patellar instability 3. D.M 4. Knee osteoarthritis 5. Previous knee surgery 6. Knee deformities involving Varus , valgus or recurvatum 7. Ligament laxity

ELIGIBILITY:
Inclusion Criteria:

* All these patients are diagnosed as lateral patellar compression syndrome depending on clinical features, MRI and diagnostic arthroscopy.

Exclusion Criteria:

1. Smoking
2. Patellar instability
3. D.M 4. Knee osteoarthritis

5. Previous knee surgery 6. Knee deformities involving Varus , valgus or recurvatum 7. Ligament laxity

Ages: 25 Years to 46 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2016-03-05 (Actual); Primary Completion 2019-11-10 (Actual); Study Completion 2019-11-25 (Actual)

PRIMARY OUTCOMES:
Lysholm knee scaling score | All patients were followed by Lysholm knee scaling score 6 months after surgery.
  Measurement of knee pain and daily activities

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hamawandi SA, Amin HI, Al-Humairi AK. Open versus arthroscopic release for lateral patellar compression syndrome: a randomized-controlled trial. Arch Orthop Trauma Surg. 2022 Oct;142(10):1-7. doi: 10.1007/s00402-021-03878-0. Epub 2021 Apr 7. PMID 33829300